CLINICAL TRIAL: NCT00611429
Title: Preparing Patients to Start Antiretroviral Therapy: A Randomized Controlled Trial
Brief Title: An Educational and Supportive Counseling Program for Increasing Antiretroviral Use and Adherence in People With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MH079700 (NIH); R01MH079700 (NIH); DAHBR 9A-ASGA
Record Dates: First submitted 2008-02-06; First posted 2008-02-11 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: HIV
Keywords: Treatment; Adherence; Intervention; Quality of Life

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Participants will receive treatment consisting of at least three individual counseling sessions and one group workshop over 12 months
  Interventions: Behavioral: Counseling sessions; Behavioral: Group workshop
- Group B (Active Comparator): Participants will receive treatment consisting of one individual counseling session and one group workshop during the last month of the study
  Interventions: Behavioral: Counseling sessions; Behavioral: Group workshop

INTERVENTIONS:
Behavioral: Counseling sessions — The individual counseling sessions will last 60 minutes and will involve discussion about health care options and information on the latest advances in HIV treatment.
Behavioral: Group workshop — During the 3-hour group workshop, doctors, nurses, and case managers will talk to participants about HIV treatments and what it is like to undergo treatment. Participants will also hear from other people with HIV and their experiences with treatment.

SUMMARY:
This study will develop and test the effectiveness of an educational and supportive counseling program called Preparing Patients to Start Antiretroviral Therapy in helping people with HIV make informed decisions about their health care.

DETAILED DESCRIPTION:
HIV is a virus that can lead to acquired immunodeficiency syndrome (AIDS), a disease that breaks down the immune system and allows for entry of life-threatening secondary infections. HIV is transmitted through the exchange of bodily fluids, primarily through sexual intercourse. Antiretroviral therapy (ART) has proven to be an effective treatment for inhibiting the replication of HIV, allowing for improved quality of life and survival.

Despite the widespread availability and effectiveness of ART, a large number of people with advanced AIDS are not on the therapy, and a number of HIV-infected people die because they are unable to access ART. The Preparing Patients to Start Antiretroviral Therapy (PATH) program is designed to inform patients about HIV treatment and to provide motivation, information, and skills to enhance treatment decision-making. The PATH program may help increase ART use and adherence. This study will develop and test the effectiveness of PATH in helping people with HIV make informed decisions about their healthcare.

This study will be divided into two phases. Phase 1 will last a total of 60 to 90 minutes and will consist of an interview about participants' relationships with friends and family and a medical history. Participants will also provide a blood sample for CD4 count and viral load measurements, returning 1 week later for the lab results. Eligible participants will then be invited to partake in Phase II of the study, which will last 12 months.

Over the 12-month study, participants in Phase 2 will be randomly assigned to Group A or Group B. Group A will be asked to attend at least three individual sessions with a counselor and one group workshop meeting with HIV experts and other people with HIV who have previously been treated with ART. The individual sessions will last 60 minutes and will involve discussion about health care options and information on the latest advances in HIV treatment. The group workshop meeting will last 3 hours and will involve teaching participants about HIV treatment and what it is like to undergo treatment. Participants assigned to Group B will attend one individual counseling session and one group workshop, both of which will cover much of the same information as the Group A sessions. Treatment for Group B will not occur until the last month of the study. Any participants in either group who decide to start taking medications for HIV during the study will be visited monthly by a research assistant who will ask about medications and check medication adherence. Participants will also be expected to check in monthly with the research team.

All participants will complete four 90-minute interviews, occurring at baseline and Months 3, 6, and 12. Interviews will include questions about relationships with friends and family, healthcare and drug-using behaviors, mental state, personal background, and education. All participants will also provide blood samples to measure CD4 count and viral load at Months 6 and 12. Selected participants may be asked to complete an additional exit interview about their opinions surrounding participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Not taking antiretroviral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2008-05; Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Treatment uptake | Measured at Month 12

SECONDARY OUTCOMES:
Treatment adherence | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Mallory O. Johnson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States